CLINICAL TRIAL: NCT05896319
Title: Hyaluronic and Synthetic Amino Acids Treatment of the Post-extraction Tooth Socket Healing in Subjects With Diabetes Mellitus Type 2: a Split-mouth Study
Brief Title: Hyaluronic Acid Treatment of the Post-extraction Tooth Socket Healing in Subjects With Diabetes Mellitus Type 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Massimo Carossa, Doctor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Unito-DM2022
Record Dates: First submitted 2023-05-02; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2; Delayed Wound Healing; Tooth Extraction Status Nos
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: split-mouth
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Postoperative application of hyaluronic acid gels 3 times per day for 7 days after tooth extraction
  Interventions: Device: Hyaluronic acid gel
- Control group (No Intervention): No adjunctive therapy undergoing natural healing

INTERVENTIONS:
Device: Hyaluronic acid gel — Post-operative application of Hyaluronic acid gel 3 times per day (8 hours distance between each application) for 7 days after oral hygiene and without swallowing, eating or drinking for one hour after the application, as follows: "wash your hands thoroughly before each application, apply a layer of gel on the injured mucosa, massage with a finger in order to facilitate spreading of the product over the treated area".
  Arms: Treatment group

SUMMARY:
The aim of the present split-mouth study was to investigate the effect of Hyaluronic Acid (HA) in improving the post-extraction tooth socket healing in subjects with diabetes mellitus type 2.

The null hypothesis was that HA can significantly improve the post extractive healing of diabetic patients compared with no treatment.

36 patients with diabetes mellitus type 2 requiring bilateral extraction of the homologous, not included, teeth were enrolled. After the extractions carried out in the same appointment, following the split-mouth design of the study, one site was randomly assigned to the test (T) group, while the other one was assigned to the control group (C).

T group included: Post-operative application of Hyaluronic acid gels 3 times per day

C group included: no treatment.

Patients were then followed after 3, 7,14 and 21 days and the healing of each socket was evaluated and compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* diabetic type 2 patients with glycaemia levels under control but with a positive history for diabetes complications (e.g., nephropathy, neuropathy, retinopathy, cardiopathy, peripheral vascular disease)
* agreement to be enrolled in the study
* availability to come at the control visit

Exclusion Criteria:

* presence of platelet dysfunction
* presence of thrombocytopenia
* corticosteroid treatment
* smokers
* refusal to participate in the study
* assumption of drugs possibly interacting with the wound healing
* extractions requiring the elevation of a flap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Change in healing index | After 3, 7, 14, and 21 days from the extraction
  3 possible scores for each of the 4 parameters considered: tissue color (1= 100% pink gum; 2=<50% hyperemic gum ; 3=>50% hyperemic gingiva), bleeding (1=absent; 2=provoked by palpation; 3=spontaneous), granulation tissue (1=pink and firm; 2=red and soft; 3=brittle), suppuration ( 1=no accumulation of plaque on the margins; 2=evident plaque on the margins; 3=suppuration/alveolitis). In this index, a score of 4 corresponds to excellent healing, conversely a score of 12 corresponds to very poor healing.
Change in residual socket volume | After 3, 7, 14, and 21 days from the extraction
  Ratio between the volume of the healing socket at a given Time and the volume of the socket at T0. It was calculated by measuring (millimeters) the maximum oral-vestibule (OV) diameter, the maximum mesio-distal (MD) diameter, and the maximum socket depth (SD). MD diameter was measured in the point of the maximum MD width of the socket both for single-rooted and multi-rooted teeth. OV diameter was measured in the point of the maximum vestibule-oral width of the socket or of each root (considering only the maximum value for the pluri-rooted teeth). SD was measured as the distance between the gingival margin and the socket bone in the point of its maximum depth (without forcing the probe).

SECONDARY OUTCOMES:
Change in pain assessment | After 3, 7, 14, and 21 days from the extraction
  Visual Analogue Scale

CONTACTS AND LOCATIONS:
Locations (1):
- C.I.R Dental School, University of Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yang S, Li Y, Liu C, Wu Y, Wan Z, Shen D. Pathogenesis and treatment of wound healing in patients with diabetes after tooth extraction. Front Endocrinol (Lausanne). 2022 Sep 23;13:949535. doi: 10.3389/fendo.2022.949535. eCollection 2022. PMID 36213270
- [Background] Marin S, Popovic-Pejicic S, Radosevic-Caric B, Trtic N, Tatic Z, Selakovic S. Hyaluronic acid treatment outcome on the post-extraction wound healing in patients with poorly controlled type 2 diabetes: A randomized controlled split-mouth study. Med Oral Patol Oral Cir Bucal. 2020 Mar 1;25(2):e154-e160. doi: 10.4317/medoral.23061. PMID 32040462
- [Background] Ibraheem W, Jedaiba WH, Alnami AM, Hussain Baiti LA, Ali Manqari SM, Bhati A, Almarghlani A, Assaggaf M. Efficacy of hyaluronic acid gel and spray in healing of extraction wound: a randomized controlled study. Eur Rev Med Pharmacol Sci. 2022 May;26(10):3444-3449. doi: 10.26355/eurrev_202205_28838. PMID 35647824
- [Background] Kim JJ, Song HY, Ben Amara H, Kyung-Rim K, Koo KT. Hyaluronic Acid Improves Bone Formation in Extraction Sockets With Chronic Pathology: A Pilot Study in Dogs. J Periodontol. 2016 Jul;87(7):790-5. doi: 10.1902/jop.2016.150707. Epub 2016 Mar 18. PMID 26991484